CLINICAL TRIAL: NCT02829801
Title: Evaluation of the Animal Intervention Used as Therapy. Impact of Animal-assisted Therapy on the Well-being in Patients With Alzheimer's Disease
Brief Title: Evaluation of the Animal Intervention Used as Therapy
Acronym: ELIAUT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 69HCL15_678
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Alzheimer Disease
Keywords: animal assisted therapy; well-being; Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AAT arm (Experimental): AAT and cognitive stimulation and rehabilitation of social tie.
  Interventions: Behavioral: AAT and cognitive stimulation and rehabilitation of social tie.
- control group (Other): Cognitive stimulation and rehabilitation of social tie.
  Interventions: Behavioral: Cognitive stimulation and rehabilitation of social tie.

INTERVENTIONS:
Behavioral: AAT and cognitive stimulation and rehabilitation of social tie. — There are 8 workshops, one workshop per week. The workshops will begin with a 15 minute introductory activity allowing the establishment of the relationship with the dog and between the participants. Activities with the dog will be offered: games, caresses, brushing.
  Then, a 40 minute cognitive stimulation will be offered. Finally, 5 minutes will be devoted to the closing of the session and to say goodbye to participants and the dog (pet him, play with him ...).
  Arms: AAT arm
Behavioral: Cognitive stimulation and rehabilitation of social tie. — There are 8 workshops, one workshop per week. The workshops will begin with an introductory activity of 15 minutes that will establish the relationship between the participants. Different topics will be proposed to foster communication and exchange.
  Then, the same cognitive stimulation in the AAT arm will be offered.
  Arms: control group

SUMMARY:
The animal-assisted therapy (AAT) is now considered a non-drug care and is often used in geriatrics. Many studies have shown a link between the presence of the animal and the psycho-behavioral symptoms decrease in dementia (PBSD) such as depression, anxiety or irritability that affects their quality of life and improved cognitive abilities. However, many methodological flaws in these researches exist.

The aim of the study is to evaluate the effectiveness of AAT on the well-being of patients with Alzheimer disease (AD) at the stage of Major Neuro Cognitive Disorder (NCD) at short and medium term (before care, during care (at the beginning and end of each session), 1 week after, 2 weeks and 1 month after the last session) compared to a group receiving the same stimulation without the dog's response.

Patients will be seen in groups of 4 to 6 people at 8 workshops. 2 groups will be formed: AAT group versus control group. The only difference between these two groups is the intervention of the dog at each workshop in the AAT group.

Each workshop will consist of three identical times. It will begin with a 15 minute introductory activity, the first goal will be to establish a relationship with patients (patients-patients and patients-caregivers) and a 40 minute cognitive stimulation, identical in the 2 groups, will be proposed and finally 5 minutes will be devoted to the closing of the session This study should highlight a positive effect of animal assisted therapy on the well-being, PBSD, depression, anxiety and cognitive abilities and a long-term retention of these positive effects.

ELIGIBILITY:
Inclusion Criteria:

Enrolled patients should have been informed and should not oppose the research, by themselves or through a trusted person, failing this, by the family, or, by a close person maintain stable ties; Subject aged over 65 years fulfilling the criteria of Alzheimer's disease the major NCD stage with or without vascular disorders; Ambulatory patient in Charpennes Day Hospital ; Being affiliated to health insurance.

Exclusion Criteria:

Patients with signs and symptoms suggestive of dementia related to other diseases than AD or mixed forms ; Patients with progressive and unstable pathologies which could interfere with the variables under consideration ; Deafness or blindness which could compromise the evaluation of the patient or his involvement during the sessions ; Patient being under guardianship ; Patient refusing the work with a animal ; Patient allergic to dogs ; Patient ending his care prior to the 13 weeks required for the study. Exclusion criteria will be sought during the questioning of the patient and his relatives as well as the review of his medical file (organic and neuroradiological explorations).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-03-02 (Actual); Primary Completion 2019-05-02 (Estimated); Study Completion 2019-05-02 (Estimated)

PRIMARY OUTCOMES:
evaluation of the changes of the well being from baseline until 3 months | before care, during care (at the beginning and end of each session), 1 week after, 2 weeks and 1 month after the last session
  Well-being will be assessed with a scale (EVIBE scale)

SECONDARY OUTCOMES:
evaluation of the changes of psycho-behavioral symptoms of dementia (PBSD) from baseline until 3 months | before and immediately after care, and 1 month after the last session.
  PBSD will be assessed by the Neuro Psychiatric Inventory, caregiver version (NPI)
evaluation of the changes of depressive symptoms from baseline until 3 months | before and immediately after care, and 1 month after the last session.
  Depressive symptoms will be measured by the Geriatric Depression Scale 30 items (GDS 30)
evaluation of the changes of the anxiety from baseline until 3 months | before and immediately after care, and 1 month after the last session.
  Anxiety will be measured by the State-Trait Anxiety Inventory (STAI)
evaluation of the changes of cognitive performances from baseline until 2 months | before et immediately after care.
  The severity of cognitive impairment will be assessed by the Alzheimer's Disease Assessment Scale, cognitive part (ADAS-Cog), GRECO version

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital des Charpennes, Villeurbanne, France